CLINICAL TRIAL: NCT03663400
Title: Identify Predictors That Distinguish Between Tofacitinib Responders and Non-responders Based on Genotype and Cellular and Molecular Profiles From Pinch Biopsies, Blood and Stool Samples
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-00630
Record Dates: First submitted 2018-08-14; First posted 2018-09-10 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Microbiota profiling by 16S sequencing RNA seq transcriptional profiling oof blood and biopsy Immunological profiling by multi parameter flow cytometry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients Treated with Tofacitinib: Microbiota profiling by 16S sequencing RNA-seq transcriptional profiling of the blood and biopsy samples Immunological profiling by multi-parameter flow cytometry
  Interventions: Diagnostic Test: GWAS analysis by Illumina BeadChip

INTERVENTIONS:
Diagnostic Test: GWAS analysis by Illumina BeadChip — will generate comprehensive genotype data for patients. Samples will be used for transcriptional profiling, microbiota profiling by 16S analysis and immunological profiling by flow cytometry

SUMMARY:
This is a prospective cohort study enrolling ulcerative colitis patients who initiate tofacitinib therapy. Investigators will collect clinical data, blood and stool samples prior to initiation of tofacitinib and, at minimum, monthly after the start of therapy. They will collect tissue from colonoscopies prior to initiation of therapy and within 6 months on therapy. Clinical characteristics and response to treatment will then be associated with genotype, blood immune profiles, stool microbiota, and cellular and molecular profiles of the biopsies to generate a treatment response model. Using predictors identified in our model, we will then attempt to validate the model and findings with the OCTAVE (Pfizer), SPARC (CCF), and RISK (CCF) data.

ELIGIBILITY:
Inclusion Criteria:

* Total mayo score between 6 and 12
* Endoscopic subscore of 2 or 3

Exclusion Criteria:

* Recent use of antibiotic therapy (<4 weeks)
* Current extreme diet (parenteral nutrition, specific carbohydrate diet).
* Active infection or malignancy.
* Significant underlying liver or renal disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18-70 with moderate to severe ulcerative colitis defined as a total mayo score between 6 and 12, and an endoscopic subscore of 2 or 3.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
GWAS analysis pretreatment | 1 Day
  GWAS analysis by Illumina BeadChip to generate comprehensive genotype data on all 50 patients.

CONTACTS AND LOCATIONS:
Overall Officials: David Hudesman, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.